CLINICAL TRIAL: NCT01499147
Title: Fludarabine Based Conditioning for Allogeneic Transplantation for Advanced Hematologic Malignancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Damiano Rondelli, MD, Professor, University of Illinois at Chicago
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000-0117
Record Dates: First submitted 2011-11-23; First posted 2011-12-26 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-10

CONDITIONS: Acute Myeloid Leukemia; Acute Leukemia; Chronic Myelogenous Leukemia; Malignant Lymphoma; Hodgkin's Disease; Multiple Myeloma; Lymphocytic Leukemia; Myeloproliferative Disorder; Polycythemia Vera; Myelofibrosis; Aplastic Anemia
Keywords: Acute myeloid leukemia; First remission; Acute lymphocytic leukemia; Acute leukemia; Second remission; Early relapse; Partial remission; Accelerated phase; Blast-crisis; Chronic myelogenous leukemia; Chronic phase; Recurrent malignant lymphoma; Refractory malignant lymphoma; Hodgkin's disease; Multiple myeloma.; Chronic lymphocytic leukemia; Myeloproliferative disorder; Polycythemia vera; Myelofibrosis; Severe aplastic anemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphoma; Hodgkin Disease; Multiple Myeloma; Leukemia, Lymphoid; Myeloproliferative Disorders; Polycythemia Vera; Primary Myelofibrosis; Anemia, Aplastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence; Blast Crisis; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — fludarabine; Busulfan; fludarabine phosphate; Melphalan; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Active Comparator): All patients below age 55 should receive fludarabine/busulfan and ATG in case of unrelated or mismatched donor.
  Interventions: Drug: fludarabine/busulfan; Drug: ATG
- Arm 2 (Active Comparator): All patients above age 55 or below age 65 should receive fludarabine/ melphalan and ATG.
  Interventions: Drug: fludarabine/ melphalan; Drug: ATG

INTERVENTIONS:
Drug: fludarabine/busulfan — All patients below age 55, should receive fludarabine/busulfan, and ATG in case of unrelated or mismatched donor, unless there is significant pulmonary, hepatic or cardiac damage: (E.g FEV1 <40%, DLCO<50%, LVEF<40, Serum bilirubin >1.5 mg% or serum transaminases > 2x nl) and/or specific medical conditions such as preventing a standard myeloablative treatment, as per discussion with the PI.
  Other Names: Fludarabine:; Fludarabine Phosphate; Fludara; Busulfan:; Busulfex; Myleran
  Arms: Arm 1
Drug: fludarabine/ melphalan — All patients above age 55 or below age 65, should receive fludarabine/melphalan, and ATG, unless there is significant pulmonary, hepatic or cardiac damage: (E.g FEV1 <40%, DLCO<50%, LVEF<40, Serum bilirubin >1.5 mg% or serum transaminases > 2x nl).
  Other Names: Fludarabine:; Fludarabine phosphate; Fludara; Melphalan:; Alkeran
  Arms: Arm 2
Drug: ATG — Patients receiving a transplant from a matched unrelated or mismatched related/unrelated donor would receive ATG in the conditioning regimen.
  Other Names: Thymoglobulin

SUMMARY:
New conditioning regimens are still needed to maximize efficacy and limit treatment-related deaths of allogeneic transplantation for advanced hematologic malignancies. Over the past several years, the investigators have evaluated several new conditioning regimens that incorporate fludarabine, a novel immunosuppressant that has limited toxicity and that has synergistic activity with alkylating agents. Recent data have suggested that fludarabine may be used in combination with standard doses of oral or IV busulfan, thus reducing the toxicity previously observed with cyclophosphamide/ busulfan regimens.

DETAILED DESCRIPTION:
Treatment-related mortality and recurrence of disease account for the majority of treatment failures in allogeneic transplantation for advanced hematologic malignancies. The most commonly utilized conditioning regimens consist of cyclophosphamide and total-body irradiation or busulfan and cyclophosphamide. Other agents such as etoposide or thiotepa are sometimes added to maximize the antileukemic effect. New conditioning regimens are however still needed to maximize efficacy and limit treatment-related deaths. Over the past several years, the investigators have evaluated several new conditioning regimens that incorporate fludarabine, a novel immunosuppressant that has limited toxicity and that has synergistic activity with alkylating agents. Recent data have suggested that fludarabine may be used in combination with standard doses of oral or IV busulfan, thus reducing the toxicity previously observed with cyclophosphamide/ busulfan regimens.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the following diseases:

  * Acute myeloid or lymphocytic leukemia in first remission at standard or high-risk for recurrence.
  * Acute leukemia in greater than or equal to second remission, or with early relapse, or partial remission.
  * Chronic myelogenous leukemia in accelerated phase or blast-crisis.
  * Chronic myelogenous leukemia in chronic phase
  * Recurrent or refractory malignant lymphoma or Hodgkin's disease
  * Multiple myeloma.
  * Chronic lymphocytic leukemia, relapsed or with poor prognostic features.
  * Myeloproliferative disorder (polycythemia vera, myelofibrosis) with poor prognostic features.
  * Severe aplastic anemia after failure of immunosuppressive therapy.
* Age 10-65 years.
* Zubrod performance status less than or equal to 2.
* Adequate cardiac and pulmonary function. Patients with decreased LVEF < 40% or DLCO < 50% of predicted will be evaluated by cardiology or pulmonary prior to enrollment on this protocol.
* Patient or guardian able to sign informed consent.

Exclusion Criteria:

* Life expectancy is severely limited by concomitant illness.
* Serum creatinine greater than 1.5 mg/dL or Creatinine Clearance less than 50 ml/min .
* Serum bilirubin greater than or equal to 2.0 mg/dl, SGPT greater than 3 x upper limit of normal
* Evidence of chronic active hepatitis or cirrhosis
* HIV-positive
* Patient is pregnant

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2000-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Damiano Rondelli, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We analyzed the clinical outcome of patients with hematological malignancies at standard or high-risk, who were transplanted (allogeneic peripheral blood or BMT HSCT) after receiving FluBU as a conditioning regimen. A total of 30 patients were recruited for this study which was conducted at the UIC Medical Center Inpatient BMT unit.
Pre-assignment Details: Criteria for FluBu conditioning: <60 years old; no diagnosis of myeloma or myelofibrosis (MF) in chronic phase; and not having received an autologous stem cell transplant with the last 2 years. Patients not fulfilling these criteria but still eligible for allogeneic transplantation were prepared with FluMel.
Groups:
- Fludarabine/Busulfan + ATG: All patients below age 55 should receive fludarabine/busulfan and ATG in case of unrelated or mismatched donor.
  fludarabine/busulfan: All patients below age 55, should receive fludarabine/busulfan, and ATG in case of unrelated or mismatched donor, unless there is significant pulmonary, hepatic or cardiac damage: (E.g FEV1 <40%, DLCO<50%, LVEF<40, Serum bilirubin >1.5 mg% or serum transaminases > 2x nl) and/or specific medical conditions such as preventing a standard myeloablative treatment, as per discussion with the PI.
- Fludarabine/Melphalan + ATG: All patients above age 55 or below age 65 should receive fludarabine/ melphalan and ATG.
  fludarabine/ melphalan: All patients above age 55 or below age 65, should receive fludarabine/melphalan, and ATG, unless there is significant pulmonary, hepatic or cardiac damage: (E.g FEV1 <40%, DLCO<50%, LVEF<40, Serum bilirubin >1.5 mg% or serum transaminases > 2x nl).
Period: Overall Study
Arm/Group | Fludarabine/Busulfan + ATG | Fludarabine/Melphalan + ATG
Started | 33 | 17
Completed | 18 | 12
Not Completed | 15 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 18 | 12 | 30
Age, Continuous [Median (Full Range); unit: years] | 34 [19 to 61] | 49 [22 to 61] | 42.5 [19 to 61]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 12 | 30
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 10 | 4 | 14
Region of Enrollment [Number; unit: participants]
  United States | 18 | 12 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Engraftment.
Description: Median time to ANC engraftment and platelet engraftment in both groups as well as the transfusion requirements measured within 30 days after transplant.
Time Frame: Up to 30 days post-transplant
Measure: Number; unit: participants
Arm/Group | Fludarabine/Busulfan + ATG | Fludarabine/Melphalan + ATG
Number analyzed (Participants) | 18 | 12
participants | 18 | 12

2. Secondary Outcome: Participants With 100 Day Transplant-related Mortality.
Description: Day 100 transplant-related mortality was measured in both groups.
Time Frame: Up to 100 days post-transplant.
Measure: Number; unit: participants
Arm/Group | Fludarabine/Busulfan + ATG | Fludarabine/Melphalan + ATG
Number analyzed (Participants) | 18 | 12
participants | 1 | 1

3. Secondary Outcome: Time to ANC and Platelet Engraftment
Description: Days to ANC or platelet engraftment
Time Frame: Up to 30 days post-transplant
Measure: Median (Full Range); unit: days to ANC and platelet engraftment
Groups:
- Fludarabine/Busulfan + ATG: All patients below age 55 should receive fludarabine/busulfan and ATG in case of unrelated or mismatched donor.
  fludarabine/busulfan: All patients below age 55, should receive fludarabine/busulfan, and ATG in case of unrelated or mismatched donor, unless there is significant pulmonary, hepatic or cardiac damage: (E.g FEV1 <40%, DLCO<50%, LVEF<40, Serum bilirubin >1.5 mg% or serum transaminases > 2x nl) and/or specific medical conditions such as preventing a standard myeloablative treatment, as per discussion with the PI.
  ATG: Patients receiving a transplant from a matched unrelated or mismatched related/unrelated donor would receive ATG in the conditioning regimen.
- Fludarabine/Melphalan + ATG: All patients above age 55 or below age 65 should receive fludarabine/ melphalan and ATG.
  fludarabine/ melphalan: All patients above age 55 or below age 65, should receive fludarabine/melphalan, and ATG, unless there is significant pulmonary, hepatic or cardiac damage: (E.g FEV1 <40%, DLCO<50%, LVEF<40, Serum bilirubin >1.5 mg% or serum transaminases > 2x nl).
  ATG: Patients receiving a transplant from a matched unrelated or mismatched related/unrelated donor would receive ATG in the conditioning regimen.
Arm/Group | Fludarabine/Busulfan + ATG | Fludarabine/Melphalan + ATG
Number analyzed (Participants) | 18 | 12
days to ANC and platelet engraftment | 15 [0 to 24] | 12 [10 to 22]

4. Secondary Outcome: Number of Participants With Moderate to Severe (Grade 2-4) Acute Graft Versus Host Disease (GVHD).
Description: Acute GVHD grade 2-4 was assessed in patients in the FluBU and FluMel groups up to 100 days after transplant.
Time Frame: Up to 100 days post-transplant (acute GVHD).
Measure: Number; unit: participants
Groups:
- Fludarabine/Melphalan +ATG: All patients above age 55 or below age 65 should receive fludarabine/ melphalan and ATG.
  fludarabine/ melphalan: All patients above age 55 or below age 65, should receive fludarabine/melphalan, and ATG, unless there is significant pulmonary, hepatic or cardiac damage: (E.g FEV1 <40%, DLCO<50%, LVEF<40, Serum bilirubin >1.5 mg% or serum transaminases > 2x nl).
Arm/Group | Fludarabine/Busulfan + ATG | Fludarabine/Melphalan +ATG
Number analyzed (Participants) | 18 | 12
participants | 2 | 1

ADVERSE EVENTS:
Time Frame: 365 days post-transplant
Description: REGIMEN-RELATED TOXICITY ACCORDING TO ORGAN SYSTEM (ref: Bearman et al: J Clin Oncol vol 6, 1988, 1562-1568)
Groups:
- Participants With Extra-hematological Toxicities: We analyzed if different rates of severe extra-hematological toxicities could be detected in patients conditioned with FluBu and FluMel and receiving PBSC.
- FluBu Participants With Extra-hematological Toxicities: We analyzed if different rates of severe extra-hematological toxicities could be detected in patients conditioned with FluBu and receiving PBSC.
- FluMel Participants With Extra-hematological Toxicities: We analyzed if different rates of severe extra-hematological toxicities could be detected in patients conditioned with FluMel and receiving PBSC.
Arm/Group | Participants With Extra-hematological Toxicities | FluBu Participants With Extra-hematological Toxicities | FluMel Participants With Extra-hematological Toxicities
Serious Adverse Events (participants affected / at risk) | 8/30 | 5/18 | 3/12
Other Adverse Events (participants affected / at risk) | 0/30 | 0/18 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Extra-hematological Toxicities (N=30) | FluBu Participants With Extra-hematological Toxicities (N=18) | FluMel Participants With Extra-hematological Toxicities (N=12)
stomatitis (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1)
CMV reactivation (Immune system disorders) | 5 (5) | 3 (3) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Extra-hematological Toxicities (N=30) | FluBu Participants With Extra-hematological Toxicities (N=18) | FluMel Participants With Extra-hematological Toxicities (N=12)
Veno-occlusive disease (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes